CLINICAL TRIAL: NCT03630458
Title: Investigating Digestive Properties of Carbohydrate-based Foods
Brief Title: Digestive Properties of Carbohydrate-based Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Distinguished Professor of Food Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1706019348
Record Dates: First submitted 2018-06-27; First posted 2018-08-14 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Appetitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pearl millet couscous - made in Senegal (Experimental): Steamed pearl millet couscous - commercially produced in Senegal
  Interventions: Other: Pearl millet couscous - made in Senegal
- Pearl millet couscous - made in USA (Experimental): Steamed pearl millet couscous - pearl millet obtained from Senegal but processed and prepared in USA
  Interventions: Other: Pearl millet couscous - made in USA
- Pearl millet thick porridge (Experimental): Thick porridge prepared according to traditional West African methods with pearl millet obtained from Senegal but processed and prepared in USA
  Interventions: Other: Pearl millet thick porridge
- Wheat couscous (Experimental): Steamed wheat couscous - wheat flour processed and prepared in USA
  Interventions: Other: Wheat couscous
- White rice (Active Comparator): White rice - medium-grain prepared using a rice cooker
  Interventions: Other: White rice

INTERVENTIONS:
Other: Pearl millet couscous - made in Senegal — Pearl millet couscous (made in Senegal) was tested for gastric emptying rate, glycemic response, fermentability, and appetitive response.
  Arms: Pearl millet couscous - made in Senegal
Other: Pearl millet couscous - made in USA — Pearl millet couscous (made in USA) was tested for gastric emptying rate, glycemic response, fermentability, and appetitive response.
  Arms: Pearl millet couscous - made in USA
Other: Pearl millet thick porridge — Pearl millet thick porridge was tested for gastric emptying rate, glycemic response, fermentability, and appetitive response.
  Arms: Pearl millet thick porridge
Other: Wheat couscous — Wheat couscous was tested for gastric emptying rate, glycemic response, fermentability, and appetitive response.
  Arms: Wheat couscous
Other: White rice — White rice was tested as a comparator for gastric emptying rate, glycemic response, fermentability, and appetitive response.
  Arms: White rice

SUMMARY:
Gastric emptying rate, glycemic response, fermentation, and appetitive response are being assessed after consumption of traditional West African carbohydrate-based foods (pearl millet couscous, pearl millet thick porridge) and Western type carbohydrate-based foods (wheat couscous, white rice).

DETAILED DESCRIPTION:
Anecdotal evidence suggests that couscous made from pearl millet (Pennisetum glaucum), hereby referred to as millet couscous, is highly satiating in populations living in the West African Sahel. Results from a previous human study conducted the investigators indicated that traditional West African foods made from pearl millet and sorghum (millet couscous, millet thick porridge, and sorghum thick porridge) exhibit markedly delayed rates of gastric emptying compared to Western foods (pasta, boiled potatoes, and white rice) in a population from Mali, Africa. The delayed gastric emptying rate of the thick porridges can be attributed at least partially to the impact of viscosity, while the cause of the delayed gastric emptying rate of the millet couscous remains unclear. The overall aim of this research is to determine why millet couscous exhibits a delayed rate of gastric emptying, while also assessing other digestive properties to gain a better understanding of the factors that could be contributing to this outcome. Therefore, gastric emptying rate, glycemic response, fermentation, and appetitive response are all being assessed for West African and Western foods in a population residing in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (18.5 < BMI < 25 kg/m2)
* Normal fasting blood glucose

Exclusion Criteria:

* Diabetes
* Allergy to millet
* Allergy or sensitivity/intolerance to gluten
* History of gastrointestinal disease
* Pregnant or nursing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | Acute study; 4 hours of measurement after consumption of test food
  Breath test is being performed using 13C-octanoic acid mixed into test meals.
Glycemic response | Acute study; 4 hours of measurement after consumption of test food
  Blood glucose is being measured using continuous glucose monitors.

SECONDARY OUTCOMES:
Breath hydrogen (fermentability) | Acute study; 4 hours of measurement after consumption of test food
  Breath samples are being collected at certain intervals for 4 hours after consumption of test food and analyzed for hydrogen levels using a breath analyzer. Breath hydrogen levels are indicative of a food's fermentability.
Appetitive response | Acute study; 4 hours of measurement after consumption of test food
  Hunger and fullness scores are being measured using a 10-cm scale (0 = weakest feeling of hunger or fullness and 10 = strongest feeling of hunger or fullness) after consumption of test food. Weaker feelings of hunger and stronger feelings of fullness are indicative of better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.